CLINICAL TRIAL: NCT00126893
Title: Phase 1 Study to Determine the Optimal Biologic Dose of CC-401 in Subjects With High-Risk Myeloid Leukemia
Brief Title: Study to Determine the Optimal Biologic Dose of CC-401 in Subjects With High-Risk Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Organization: Celgene (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-401-AML-001
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2006-12

CONDITIONS: Myeloid Leukemia
Keywords: Leukemia; AML; CC401; CC-401; Celgene; High Risk Myeloid Leukemia; Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia | interventions — CC 401

INTERVENTIONS:
Drug: CC-401

SUMMARY:
This is a single center Phase 1 study to evaluate the safety, pharmacokinetics and pharmacodynamics of CC-401 in subjects with refractory acute myelogenous leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form.
* Must be greater than or equal to 18 years of age at the time of signing the informed consent form.
* Must have a diagnosis of high-risk myeloid leukemia, defined as:

  1. Subjects > 70 years of age with newly diagnosed acute myelogenous leukemia (AML) (regardless of karyotype) who decline conventional induction chemotherapy;
  2. Subjects > 60 years of age with newly diagnosed AML and poor-risk cytogenetics or a history of secondary AML who decline conventional induction chemotherapy;
  3. Subjects with newly diagnosed AML who do not experience a CR after at least 2 cycles of induction chemotherapy;
  4. Subjects with AML who do not experience a second or greater complete remission after 1 but no more than 2 cycles of re-induction chemotherapy;
  5. Subjects with recurrence of AML after a remission duration of less than three months in subjects < 60 years of age or remission duration of less than six months in subjects > 60 years of age; or
  6. Subjects with imatinib-refractory chronic myeloid leukemia (CML) in blast crisis defined as > 30% blasts and promyelocytes in the peripheral blood or bone marrow smear despite treatment with imatinib > 600 mg/daily
* ECOG performance status < 2 (see Appendix 2).
* Serum creatinine < 2 mg/d and ALT (SGPT), alkaline phosphatase, and conjugated bilirubin < 2 times the upper limit of normal.
* No conventional or investigational anti-leukemic treatment within two weeks of the administration of study drug with the exception of hydroxyurea to control the peripheral blood blast count.
* Subjects must have recovered from any prior treatment-related toxicities.
* Subject must be able to adhere to the study visit schedule and other protocol requirements.
* Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days of starting study drug. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study drug. WCBP must agree to have pregnancy tests every 4 weeks while on study drug.
* Males (including those who have had a vasectomy) must use barrier contraception (latex condoms) when engaging in reproductive sexual activity with WCBP while on study medication and 4 weeks after the last dose of study medication

Exclusion Criteria:

* Subjects with central nervous system (CNS) involvement as documented by spinal fluid cytology or imaging; individuals with signs or symptoms of leukemic meningitis or a history of leukemic meningitis must have a negative lumbar puncture within 2 weeks prior to enrollment in the study.
* Subjects who are pregnant or lactating; women of child-bearing potential must have a negative urine or serum pregnancy test within 14 days prior to the initial treatment with CC-401.
* Subjects with severe or life threatening active, unresolved systemic infections.
* Prior history of malignancy other than myeloid leukemia (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for ≥ 3 years.
* Known HIV-1 positivity.
* Known hepatitis B surface antigen (HBsAg) positivity.
* Prior treatment with CC-401
* Use of any other experimental drug or treatment within 28 days of baseline
* Inability to provide a bone marrow aspirate
* Subjects with severe or life-threatening active bleeding refractory to platelet transfusion
* Subjects with severe or life-threatening anemia refractory to red blood cell transfusion
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2005-10; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Medical Center, Indianapolis, Indiana, United States